CLINICAL TRIAL: NCT05294315
Title: The Analgesic Efficacy of Bi-level Versus Single Level Erector Spinae Block in Video Assisted Thoracoscopic Surgery: a Randomized Patient Blinded Study
Brief Title: Bi-level vs. Single Level ESB in VATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Cheng Lin, Clinical Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 120374
Record Dates: First submitted 2022-01-11; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single level block arm - Control (Active Comparator): Single level erector spinae block at 4th transverse process
  Interventions: Procedure: Single level erector spinae block
- Bi-level block arm - Intervention (Experimental): Bi-level erector spinae block at 4th and 6th transverse process
  Interventions: Procedure: Bi-level erector spinae block

INTERVENTIONS:
Procedure: Bi-level erector spinae block — erector spinae block at 4th and 6th transverse process
  Arms: Bi-level block arm - Intervention
Procedure: Single level erector spinae block — erector spinae block at 4th transverse process
  Arms: Single level block arm - Control

SUMMARY:
Video assisted thoracoscopic surgery (VATS) is a minimally invasive surgery to remove lesions from the thoracic cavity. It is associated with moderate pain which can lead to pulmonary complications after surgery. The Enhanced Recovery After Surgery (ERAS) and the European Society of Thoracic Surgeons recommended a multimodal analgesia approach to manage pain after VATS. Erector spinae block (ESB) is a popular analgesic block due to its ease of performance and wide coverage. It has been shown to be effective in randomized control trials. Recently, case reports on bi-level ESB are emerging, suggesting more effective analgesia compared to single level ESB. As there is no available data, the investigators are interested in conducting a randomized pilot study, comparing bi-level to single level ESB to gather baseline data for sample size calculation for a formal randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (at least 18 years old)
* elective unilateral wedge resection, segmentectomy, lobectomy or bilobectomy via VATS

Exclusion Criteria:

* history of malignant hyperthermia
* BMI > 40, chronic pain condition
* Daily opioid consumption of more than 60 mg oral morphine equivalents
* Conversion to thoracotomy
* Insertion of epidural
* postoperative admission to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Opioid use in first 12 postoperaive hour | First 12 hour from arriving at postoperative recovery

SECONDARY OUTCOMES:
Pain score area under curve first 12 hour | First 12 hour from arriving at postoperative recovery
  Numeric rating scale, 0 to 10, 0 being no pain and 10 being the worst possible pain
Pain score area under curve first 24 hour | First 24 hour from arriving at postoperative recovery
  Numeric rating scale, 0 to 10, 0 being no pain and 10 being the worst possible pain
Incidence of Acute block complication - based on clinical assessment | First 12 hour since block placement
  pneumothorax, local anesthetic toxicity, epidural spread, bleeding
Incidence of Delayed block complication - based on clinical assessment | First 5 days
  paresthesia, motor weakness, hematoma, abscess

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Lin, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided